CLINICAL TRIAL: NCT04627038
Title: Randomized, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate LY3556050 for the Treatment of Osteoarthritis Pain
Brief Title: Chronic Pain Master Protocol (CPMP): A Study of LY3556050 in Participants With Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17593; H0P-MC-OA03 (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3556050 600 mg (Experimental): Participants received 600 mg LY3556050 twice daily (BID) every 12 hours for up to 8 weeks.
  Interventions: Drug: LY3556050
- Placebo (Placebo Comparator): Participants received placebo BID every 12 hours for up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3556050 — LY3556050 Given orally
  Arms: LY3556050 600 mg
Drug: Placebo — Placebo Given orally
  Arms: Placebo

SUMMARY:
This study is being done to test the safety and efficacy of LY3556050 for the treatment of osteoarthritis pain. This trial is part of the chronic pain master protocol, H0P-MC-CPMP (NCT05986292), which is a protocol to accelerate the development of new treatments for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a visual analog scale (VAS) pain value ≥40 and <95 during screening.
* Have a history of daily pain for at least 12 weeks based on participant report or medical history.
* Have a body mass index <40 kilograms per meter squared (kg/m²) (inclusive).
* Are willing to maintain a consistent regimen of any ongoing nonpharmacologic pain-relieving therapies (for example, physical therapy) and will not start any new nonpharmacologic pain-relieving therapies during study participation.
* Are willing to discontinue all medications taken for chronic pain conditions for the duration of the study.
* Have presence of index knee pain for >12 weeks at screening.
* Have an x-ray supporting diagnosis of osteoarthritis according to the American College of Rheumatology with a Kellgren-Lawrence grade 2 to 4 radiographic classification of index knee.
* Are men, or women able to abide by reproductive and contraceptive requirements.

Exclusion Criteria:

* Have second- or third-degree atrioventricular (AV) heart block or AV dissociation or history of ventricular tachycardia.
* Have had a procedure within the past 6 months intended to produce permanent sensory loss in the target area of interest (for example, ablation techniques).
* Have surgery planned during the study for any reason, related or not to the disease state under evaluation.
* Have, in the judgment of the investigator, an acute, serious, or unstable medical condition or a history or presence of any other medical illness that would preclude study participation.
* Have had cancer within 2 years of baseline, except for cutaneous basal cell or squamous cell carcinoma resolved by excision.
* Have a substance use disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (5th edition; DSM-5; American Psychiatric Association).
* Have a positive human immunodeficiency virus (HIV) test result at screening.
* Are in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Have an intolerance to acetaminophen or paracetamol or any of its excipients.
* Have a history of alcohol, illicit drug, analgesic or narcotic use disorder within 2 years prior to screening.
* Are largely or wholly incapacitated and unable to participate fully in all protocol procedures, for example, bedridden or confined to a wheelchair, permitting little or no selfcare.
* Have presence of surgical hardware or other foreign body in the index knee.
* Have an unstable index joint (such as a torn anterior cruciate ligament).
* Have had a surgical procedure or therapeutic injection in the affected knee within 3 months prior to starting the washout period.
* Have fibromyalgia, chronic pain syndrome, or other concurrent medical or arthritic conditions that could interfere with the evaluation of the index knee.
* Have a history of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis, or amyloidosis.
* Have clinical signs and symptoms of active knee infection or crystal disease of the index knee.
* Have a history of infection in the index joint.
* Have a history of arthritis due to crystals (e.g., gout, pseudogout).
* Have pain or functional impairment due to ipsilateral hip osteoarthritis.
* Have a history within 2 years prior to screening or current evidence of syncope, presyncope, uncontrolled vertigo, or postural dizziness, judged to be clinically significant by the investigator.
* Have clinically significant active thyroid disease, including Hashimoto's thyroiditis.
* Are taking metformin therapy.
* Are pregnant or breastfeeding.
* Have had any joint replacement such as knee of the lower extremity, such as hip, knee or ankle, in the past 6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (38):
  - Simon Williamson Clinic, Birmingham, Alabama
  - Synexus- Chandler, Chandler, Arizona
  - Synexus Clinical Research - Glendale, Glendale, Arizona
  - Alliance for Multispecialty Research - Clinical Research Consortium, Tempe, Arizona
  - Irvine Clinical Research, Irvine, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - CMR of Greater New Haven, Hamden, Connecticut
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Suncoast Research Group, Miami, Florida
  - University of Miami Don Suffer Clinical Research Building, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Synexus Clinical Research US, Inc - Orlando, Orlando, Florida
  - Synexus Clinical Research - St. Petersburg, Pinellas Park, Florida
  - Martin E. Hale M.D., P.A., Plantation, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Synexus Clinical Research, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices and Research, Methuen, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - PharmQuest, Greensboro, North Carolina
  - Synexus - Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Clinical Research Center of Reading,LLC, Wyomissing, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Cedar Health Research, Dallas, Texas
  - Synexus - US, San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Puerto Rico (2):
  - Ponce Medical School Foundation Inc., Ponce
  - Latin Clinical Trial Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Chronic Pain Master Protocol (CPMP): A Study of LY3556050 in Participants With Osteoarthritis — https://trials.lillytrialguide.com/en-US/trial/3dzoGaeE7LytIIXgbs84eS

RESULTS

PARTICIPANT FLOW:
Groups:
- LY3556050 600 Milligram (mg): Participants received 600 mg LY3556050 twice daily (BID) every 12 hours for up to 8 weeks.
Period: Overall Study
Arm/Group | LY3556050 600 Milligram (mg) | Placebo
Started | 135 | 67
Received at Least One Dose of Study Drug | 135 | 66
Completed | 81 | 53
Not Completed | 54 | 14
Not completed — Adverse Event | 36 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 13 | 3
Not completed — Non-compliance with study drug | 0 | 1
Not completed — Prohibited Concomitant Medication | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- LY3556050 600 mg: Participants received 600 mg LY3556050 BID every 12 hours for up to 8 weeks.
- Total: Total of all reporting groups
Arm/Group | LY3556050 600 mg | Placebo | Total
Number analyzed (Participants) | 135 | 67 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 33 | 109
  >=65 years | 59 | 34 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.4) | 62.8 (8.8) | 62.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 39 | 116
  Male | 58 | 28 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 10 | 37
  Not Hispanic or Latino | 108 | 57 | 165
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 13 | 36
  White | 106 | 51 | 157
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 135 | 67 | 202
Average Pain Intensity as Measured by the Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: score on a scale] — The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  score on a scale | 5.58 (1.68) | 5.54 (1.57) | 5.57 (1.64)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Pain Intensity as Measured by the Numeric Rating Scale (NRS)
Description: The NRS was used to describe pain severity. Participants were asked to describe their average pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  Posterior mean change from baseline, 95 percent (%) credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: All enrolled participants who received at least one dose of study drug. Here, the overall number of participants analyzed includes the number of participants with non-missing value at Week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 63 | 46
score on a scale | -1.67 [-2.05 to -1.30] | -1.76 [-2.23 to -1.29]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.09, 95% CI 2-sided [-0.51 to 0.67] — Posterior mean difference with 95% credible interval is reported

2. Secondary Outcome: Change From Baseline on the Western Ontario and McMaster University Arthritis Index (WOMAC®) Pain Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 5 questions on the pain subscale, and participants used a 0 to 4 Likert scale to answer each question for the current day: 0 = no pain, and 4 = extreme pain. The scores for the pain subscale were calculated by summing the scores of the 5 questions for each participant at each time point. The range of possible scores is 0 to 20 with higher scores representing worse outcome.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 81 | 53
score on a scale | -2.57 [-3.22 to -1.90] | -3.51 [-4.35 to -2.67]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.95, 95% CI 2-sided [-0.07 to 1.96] — Posterior mean difference with 95% credible interval is reported

3. Secondary Outcome: Change From Baseline on the WOMAC® Stiffness Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 2 questions in the stiffness subscale and participants used a 0 to 4 Likert scale to answer each question for the current day: 0 = no stiffness, and 4 = extreme stiffness. The scores for the stiffness subscale was calculated by summing the scores of the 2 questions for each participant at each time point. The range of possible scores is 0 to 8 with higher scores representing worse outcome.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 81 | 53
score on a scale | -1.15 [-1.48 to -0.81] | -1.39 [-1.79 to -0.99]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.24, 95% CI 2-sided [-0.24 to 0.72] — Posterior mean difference with 95% credible interval is reported

4. Secondary Outcome: Change From Baseline on the WOMAC® Physical Function Subscale
Description: The WOMAC® is a validated instrument that is extensively used to evaluate the response to medications for the treatment of Osteoarthritis pain. There are 17 questions in the physical function subscale, and participants used a 0 to 4 Likert scale to answer each question for the current day: 0 = no difficulty, and 4 = extreme difficulty. The score for physical function subscale was calculated by summing the scores of the 17 questions for each participant at each time point. The range of possible scores is 0 to 68 with higher scores representing worse outcome.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 81 | 53
score on a scale | -8.33 [-10.45 to -6.17] | -12.18 [-14.92 to -9.39]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = 3.84, 95% CI 2-sided [0.39 to 7.20] — Posterior mean difference with 95% credible interval is reported

5. Secondary Outcome: Change From Baseline for Overall Improvement as Measured by Patient's Global Impression of Change
Description: Patients Global Impression of Change captured the participant's perspective of treatment apart from sub-aspects of the general improvement. This is a numeric scale from 1 to 7: 1 = very much better, and 7 = very much worse.
  Posterior mean, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 81 | 53
score on a scale | 2.76 [2.53 to 3.00] | 2.86 [2.57 to 3.16]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.10, 95% CI 2-sided [-0.48 to 0.28] — Posterior mean difference with 95% credible interval is reported

6. Secondary Outcome: Change From Baseline for Worst Pain Intensity as Measured by NRS
Description: The NRS was used to describe pain severity. Participants were asked to describe their worst pain over the past 24 hours, on a scale of 0 to 10: 0 = no pain, and 10 = pain as bad as you can imagine.
  Posterior mean, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 63 | 46
score on a scale | -1.74 [-2.14 to -1.33] | -2.05 [-2.55 to -1.54]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.31, 95% CI 2-sided [-0.32 to 0.95] — Posterior mean difference with 95% credible interval is reported

7. Secondary Outcome: Change From Baseline on the Visual Analog Scale (VAS) for Pain
Description: VAS was a graphic, single-item scale where participants were asked to describe their pain intensity over the past week, on a scale of 0 to 100: 0 = no pain, and 100 = worst imaginable pain. Participants completed the VAS by placing a line perpendicular to the VAS line at a point that described their pain intensity.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 81 | 53
score on a scale | -19.69 [-24.36 to -15.05] | -25.93 [-31.84 to -19.93]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = 6.24, 95% CI 2-sided [-1.05 to 13.56] — Posterior mean difference with 95% credible interval is reported

8. Secondary Outcome: Change From Baseline on the Sleep Scale From the Medical Outcomes Study (MOS Sleep Scale) - Average Hours of Sleep
Description: The MOS Sleep Scale consists of 12 questions addressing the past week. Question 1 asks time to fall asleep and it is reported in 5-point timeframe categories. Question 2 asks average hours of sleep. In the remaining 10 questions participants report how often a sleep symptom or problem was present on a scale ranging from '0=all of the time' to '5=none of the time.' MOS Sleep scale dimension scores range from 0 to 100 with lower score indicating improvement, except for the dimension of sleep adequacy, where higher scores indicate improvement. Here, the average hours of sleep (i.e., Question 2) is reported as the average number of hours slept each night during the past week (range 0 to 24 hours). Higher number of hours slept indicates improvement.
  Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Hours per night
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 81 | 52
Hours per night | 0.15 [-0.05 to 0.34] | -0.01 [-0.25 to 0.23]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = 0.16, 95% CI 2-sided [-0.14 to 0.46] — Posterior mean difference with 95% credible interval is reported

9. Secondary Outcome: Total Amount of Rescue Medication Use as Measured by Average Daily Dosage
Description: Total amount of rescue medication use as measured by average daily dosage. Posterior mean change from baseline, 95% credible interval was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg per day (mg/day)
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 63 | 46
mg per day (mg/day) | 247.24 [146.10 to 349.69] | 248.06 [115.23 to 380.78]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.82, 95% CI 2-sided [-166.74 to 165.52] — Posterior mean difference with 95% credible interval is reported

10. Secondary Outcome: Change From Baseline on the EuroQuality of Life Five Dimensions (5D) Five Level (5L) Questionnaire (EQ-5D-5L) Health State Index (United States Algorithm)
Description: The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension. The scores in the 5 dimensions were summarized into a health state index score using the United States algorithm. The health state index value is a single value on a scale from less than 0 to 1 (negative values are valued as worse than dead) with higher scores indicating better health: 0=a health state equivalent to death, and 1=perfect health.
  Posterior mean change from baseline, 95% credible intervals was derived using Bayesian mixed model repeated measures. Data presented are posterior mean with 95% credible interval.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | LY3556050 600 mg | Placebo
Number analyzed (Participants) | 81 | 53
score on a scale | 0.03 [-0.02 to 0.09] | 0.05 [-0.01 to 0.11]
Statistical Analysis 1: Comparison: LY3556050 600 mg vs Placebo; Test type: Superiority; Posterior Mean Difference = -0.02, 95% CI 2-sided [-0.09 to 0.06] — Posterior mean difference with 95% credible interval is reported

ADVERSE EVENTS:
Time Frame: Baseline through Week 8
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | LY3556050 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/135 | 2/66
Other Adverse Events (participants affected / at risk) | 83/135 | 24/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3556050 600 mg (N=135) | Placebo (N=66)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3556050 600 mg (N=135) | Placebo (N=66)
Abdominal discomfort (Gastrointestinal disorders) | 7 (8) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 8 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 29 (31) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 26 (29) | 6 (8)
Fatigue (General disorders) | 19 (21) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (9)
Dizziness (Nervous system disorders) | 22 (25) | 1 (2)
Headache (Nervous system disorders) | 8 (8) | 7 (12)
Lethargy (Nervous system disorders) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT04627038/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT04627038/SAP_001.pdf